CLINICAL TRIAL: NCT01491074
Title: Effect of the Interleukin-6 Receptor Antagonist Tocilizumab in Non-ST Elevation Myocardial Infarction - a Randomized, Double Blind, Placebo Controlled Study.
Brief Title: Effect of the Interleukin-6 Receptor Antagonist Tocilizumab in Non-ST Elevation Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010/1971 [REK]; 2010-021953-37 (EudraCT Number); 2010/1971 (Registry Identifier: REK); 10/15070-4 (Registry Identifier: SLV); 4947 (Other Grant/Funding Number: HSØ); 2010/19043 (Other: PVO)
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Non-ST Elevation Myocardial Infarction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NaCl 0.9% 100 ml (Placebo Comparator)
  Interventions: Drug: NaCl 0.9% 100 ml
- Tocilizumab 280 mg (Experimental): Intravenous infusion, 280 mg Tocilizumab (14 ml) added to 86 ml of 0.9% NaCl
  Interventions: Drug: Tocilizumab 280 mg

INTERVENTIONS:
Drug: Tocilizumab 280 mg — Intravenous administration of 280 mg Tocilizumab (14 ml), mixed with 86 ml 0.9% NaCl
  Other Names: Brand name RoActemra (Roche); ATC: L04A C07
  Arms: Tocilizumab 280 mg
Drug: NaCl 0.9% 100 ml — Placebo
  Arms: NaCl 0.9% 100 ml

SUMMARY:
Acute coronary syndromes (ACS) are still associated with high morbidity and mortality, despite several improvements in their management. This may indicate that important pathogenic mechanisms contribute to both stable and unstable atherosclerotic disease mechanisms.

Based upon previous research, the investigators believe that providing a block in the damaging inflammatory loop though short term inhibition of Interleukin-6 receptor signalling, could be an attractive therapeutic target in ACS; and of particular interest in patients with non-ST elevation myocardial infarction (NSTEMI), a disease often characterized by widespread coronary inflammation with multiple unstable plaques.

The investigators hypothesize that a single administration of the anti-Interleukin 6 receptor antagonist Tocilizumab, in patients with NSTEMI, may interrupt the self-perpetuating inflammatory loops which could improve plaque stability, with potential secondary beneficial effects on myocardial damage.

This will be investigated in a randomized, double blind, placebo-controlled study, including a total of 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* NSTEMI (ESC Type 1)
* Age 18-80 years
* Troponin T >/= 30 ng/ml
* Informed consent to participation

Exclusion Criteria:

* STEMI
* Known cardiac disease, except coronary disease (cardiomyopathy, heart failure with known EF < 45%, severe valvular heart disease attending regular follow-up, recent PCI/ACB (< 3 months))
* Hemodynamic and/or respiratory instability
* Cardiac arrest in acute phase
* Concurrent condition affecting/potentially affecting CRP (infection, malignancy, autoimmune disease)
* Recent major surgery (< 3 months)
* Recent/concurrent immunosuppressant treatment (< 2 weeks, except NSAIDs)
* Severe renal failure (eGFR < 30 ml/min)
* Pregnancy
* Contraindications to any study investigations and/or medication.
* Expected non-adherence to study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
high sensitivity C-reactive protein Area under the curve (AUC) | 0-56 hrs following inclusion

SECONDARY OUTCOMES:
hs troponin T | 0-56 hrs, 3 months and 6 months following inclusion
hs CRP | 3 and 6 months following inclusion
pro-BNP | 0-56 hrs, 3 and 6 months
Infarct size | 6 months
  Assessed by Echocardiography and MRI at 6 months
LV size | acute phase (0-3 days), 6 months
  Assessed by echocardiography
LV function | acute phase (0-3 days), 6 months
  Assessed by echocardiography, cardiac MRI at 6 months
Coronary flow reserve | acute phase (0-3 days), 6 months
  Assesses coronary microvascular function - for 60 patients only.
Endothelial function | Acute phase (0-3 days) and 6 months
  Assessed by tonometry

OTHER OUTCOMES:
Other inflammatory pathways | 0-56 hrs, 3 monhts, 6 months
  TNF-alfa, IL-1, IL-6, IL-18, platelet-derived inflammatory mediators, anti-inflammatory cytokines etc

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, MD, PhD, Principal Investigator — Oslo University Hospital; Rune Wiseth, MD, PhD, Study Chair — St. Olavs Hospital; Pål Aukrust, MD, PhD, Study Chair — Oslo University Hospital; Jan K Damås, MD, PhD, Study Chair — St. Olavs Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo, Oslo County
  - St Olavs Hospital, Trondheim, Sør-Trøndelag

REFERENCES:
- [Derived] Aherrahrou R, Reinberger T, Hashmi S, Erdmann J. GWAS breakthroughs: mapping the journey from one locus to 393 significant coronary artery disease associations. Cardiovasc Res. 2024 Nov 5;120(13):1508-1530. doi: 10.1093/cvr/cvae161. PMID 39073758
- [Derived] Ueland T, Kleveland O, Michelsen AE, Wiseth R, Damas JK, Aukrust P, Gullestad L, Halvorsen B, Yndestad A. Serum PCSK9 is modified by interleukin-6 receptor antagonism in patients with hypercholesterolaemia following non-ST-elevation myocardial infarction. Open Heart. 2018 Sep 18;5(2):e000765. doi: 10.1136/openhrt-2017-000765. eCollection 2018. PMID 30258647
- [Derived] Kleveland O, Ueland T, Kunszt G, Bratlie M, Yndestad A, Broch K, Holte E, Ryan L, Amundsen BH, Bendz B, Aakhus S, Espevik T, Halvorsen B, Mollnes TE, Wiseth R, Gullestad L, Aukrust P, Damas JK. Interleukin-6 receptor inhibition with tocilizumab induces a selective and substantial increase in plasma IP-10 and MIP-1beta in non-ST-elevation myocardial infarction. Int J Cardiol. 2018 Nov 15;271:1-7. doi: 10.1016/j.ijcard.2018.04.136. Epub 2018 Jun 29. PMID 29961572